CLINICAL TRIAL: NCT02467140
Title: A Clinical Study of Postoperative Pain Following Laparoscopic Transabdominal Preperitoneal Inguinal Hernioplasty. Comparing Parietex ProGrib With Tacks for Mesh Fixation
Brief Title: Comparing Pain After Laparoscopic Hernia Repair Using Two Different Types of Mesh Fixation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2307PG
Record Dates: First submitted 2015-06-04; First posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-05

CONDITIONS: Inguinal Hernia; Pain
Keywords: Inguinal hernia repair; Hernia; ProGrib self-fixating mesh; Biological mesh; Tack fixation
MeSH Terms: conditions — Hernia, Inguinal; Pain; Hernia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-fixating mesh (Active Comparator): During surgery, the Parietex ProGrib mesh will be used.
  Interventions: Device: Parietex ProGrib self-fixating mesh
- Tack fixation (Active Comparator): During surgery, the mesh will be fixated with tacks.
  Interventions: Device: Tack fixation

INTERVENTIONS:
Device: Parietex ProGrib self-fixating mesh — Laparoscopic transabdominal preperitoneal inguinal hernioplasty using the Parietex ProGrib self-fixating mesh.
  Arms: Self-fixating mesh
Device: Tack fixation — Laparoscopic transabdominal preperitoneal inguinal hernioplasty using the Parietex ProGrib self-fixating mesh using tack fixation.
  Arms: Tack fixation

SUMMARY:
A clinical study evaluating acute and chronic pain following laparoscopic inguinal hernia repair comparing the ProGripTM self- fixating mesh with tack fixation.

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate acute and chronic pain following laparoscopic inguinal hernia repair comparing the ProGripTM self- fixating mesh with tack fixation. The ProGripTM laparoscopic self-fixating mesh has been approved for implantation to reinforce the abdominal wall during laparoscopic inguinal hernia repair (TAPP). The mesh delivers tack free fixation above and below the inguinal ligament potentially eliminating pain associated with traditional tack fixation. The present study is a prospective randomized clinical trial designed to collect information about complications such as acute and chronic pain and hernia recurrence rate from patients referred for laparoscopic inguinal hernia repair. Patients who qualify to take part in the study will be randomized for a procedure using either a self-gripping ProGrip mesh or a conventional polypropylene mesh attached with AbsorbaTackTM. Data will be collected from operations performed at 6 high volume hernia centers in Denmark.

Patients eligible for study will be recruited from the referral list for inguinal hernia repair at each participating institution. Prior to scheduled surgery, patients will be consented and will complete a questionnaire on inguinal pain intensity and quality of life .

The mesh will be placed intraperitoneally after the component separation is complete. The peritoneal layer will be closed with a V-loc stitch in both groups.

After surgery, key clinical data will be recorded, such as type of mesh used, size of the hernia defect, number of tacks used etc.

The participating patients will receive postoperative questionnaires following the first year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective, inguinal hernia repair
* 18 years or older
* Male gender
* ASA physical classification system 1-3
* Informed consent

Exclusion Criteria:

* Patients with recurrent hernia, except patients operated in childhood without mesh application.
* Patients with bilateral hernia
* Patients with chronic pain
* Patients in anticoagulation therapy
* Previous major surgery in lower abdomen

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients experiencing acute postoperative pain, using the NRS pain score. | 3 months
Number of patients with recurrent hernia. | 1 year

SECONDARY OUTCOMES:
Number of patients experiencing chronic postoperative pain, using the NRS pain score. | 1 year
Quality of life before and after surgery, using the Carolina Comfort Scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Nielsen, MD PhD, Study Director
Locations (1):
- Hospitalsenheden Midt, Viborg, Region Midt, Denmark